CLINICAL TRIAL: NCT06539845
Title: Development and Effectiveness of a New Intervention on Household Preparedness for Disease X and Outbreaks Among Orang Asli in Selangor: A Cluster Randomized Trial
Brief Title: Creating a New Health Promotion Module to Help the Indigenous People of Selangor Prepare for Disease X and Outbreaks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Collaborators: Ministry of Health, Malaysia (Other Government); Universiti Putra Malaysia (Other); Institute for Health Behavioural Research (Unknown); Department of Orang Asli Development (Unknown)
Responsible Party: Principal Investigator, Ameerah Su'ad binti Abdul Shakor, Principal Investigator, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-01859-NQ7
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Attitude to Health; Behavior, Health; Health Behavior; Health-Related Behavior; Health Attitude; Health Knowledge, Attitudes, Practice; Knowledge, Attitudes, Practice; Preparedness; Outbreaks
Keywords: Indigenous People; Aboriginal; Preparedness; Readiness; Community Trial; Outbreak
MeSH Terms: conditions — Health Behavior; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Randomly selected Orang Asli villages will receive the intervention package along with educational brochures, through a workshop they will need to participate in once.
  Interventions: Behavioral: Outbreak Preparedness Intervention for the Orang Asli
- Control (Active Comparator): Randomly selected Orang Asli villages that will receive the educational brochures only.
  Interventions: Behavioral: Educational Brochures for the Orang Asli

INTERVENTIONS:
Behavioral: Outbreak Preparedness Intervention for the Orang Asli — The chosen villages will be given the intervention package, which includes a workshop, simulation exercises, and a card game, in addition to educational brochures on communicable disease prevention sourced from the Ministry of Health Malaysia "Info Sihat" website. This entire package will be delivered once, during the workshop, after they have answered the survey at T0.
  Arms: Intervention
Behavioral: Educational Brochures for the Orang Asli — The chosen villages will be given educational brochures on communicable disease prevention sourced from the Ministry of Health Malaysia "Info Sihat" website. This will be given once during the first encounter with the participant, after they have answered the survey at T0.
  Arms: Control

SUMMARY:
The goal of this cluster randomized trial is to develop and test a new method for preparing indigenous (locally termed as Orang Asli) households in Selangor, a state in Malaysia, for outbreaks and Disease X, a potential unknown infectious threat. It aims to determine if the new method, a health education package comprised of workshops, simulation exercises, and card game play sessions, can enhance the readiness of these families for such outbreaks.

The main questions it is looking to answer are:

1. Will the intervention package increase the level of preparedness for a Disease X and outbreaks among indigenous households in Selangor?
2. Will the intervention improve the awareness and attitudes of the indigenous people in Selangor towards outbreak preparedness?
3. Will it lead to more proactive preparedness actions by these households?

To evaluate the effectiveness of the intervention package, researchers will compare outcomes between two groups: the intervention group receiving both the intervention package and educational brochures on communicable disease prevention, and the control group receiving only the brochures.

Participants will:

1. Participate in the activities in the newly developed intervention package, which would include workshops, simulation exercises, and card game play sessions.
2. Answer surveys four times: before, immediately after, 1 month after and 2 months after the intervention, to measure any changes in their preparedness levels for an outbreak.

ELIGIBILITY:
Inclusion Criteria:

* Orang Asli ethnicity
* Malaysian citizen
* Age between 18 to 99 years old
* The head of the household, or the person who contributes to, or influences health-related decisions for the household
* Live in a household with at least three members
* Able to converse in Malay

Exclusion Criteria:

* Having physical or cognitive disabilities (e.g., blindness, deafness, schizophrenia and dementia)
* Having severe health conditions (e.g., respiratory and cardiovascular disease requiring oxygen support such as severe asthma/chronic obstructive pulmonary disease/heart failure and congenital heart diseases)
* Residing temporarily (less than 2 years)
* Intending to relocate to a different residence within the next 2 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Household Preparedness Score | Before intervention (T0), immediately after the intervention (T1), 1-month follow-up (T2), and at a 2-months follow-up (T3)
  The combined scores of awareness/attitude and the preparedness actions of the participant in a specific area towards potential disasters. The preparedness level is measured on a 4-category scale: Fully prepared, Committed, Aware, and Least prepared or unprepared.
Household Preparedness Matrix | Before intervention (T0), immediately after the intervention (T1), 1-month follow-up (T2), and at a 2-months follow-up (T3)
  Based on the "Household Preparedness Score", the level of preparedness by assigning each respondent a position on the matrix based on their questionnaire responses.

SECONDARY OUTCOMES:
Cognitive Preparedness score | Before intervention (T0), immediately after the intervention (T1), 1-month follow-up (T2), and at a 2-months follow-up (T3)
  Measures the knowledge and attitude of participant regarding outbreak and Disease X awareness Additionally, gathering insights about people's perception of possible risk hazard that may affect them including the consequences and how to mitigate. The score is derived from the total sum of marks gathered from each item within the Knowledge and Attitude domain and normalized into a scale of 0 to 1.
Preparedness Behaviour score | Before intervention (T0), immediately after the intervention (T1), 1-month follow-up (T2), and at a 2-months follow-up (T3)
  Measures the current level of preparedness actions that has been done by participants. The score is derived from the total sum of marks gathered from each item within the Practice domain and normalized into a scale of 0 to 1.

CONTACTS AND LOCATIONS:
Overall Officials: Ameerah Su'ad Abdul Shakor, Principal Investigator — Universiti Teknologi Mara
Locations (1):
- Pejabat JAKOA Daerah Gombak dan Petaling, Gombak, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the published study results may be considered for sharing but will not be distributed without the consent of Universiti Teknologi Mara, the Ministry of Health Malaysia, and the Department of Orang Asli Development. Other researchers must first obtain permission from these entities. The datasets generated or analyzed during this study will not contain any identifiers and will be made available to other researchers upon request after receiving their approval. The decision regarding the extent of data to be shared will be based on the reasonableness of the request. Participants can request access to their own individual results but not to those of other participants. Additionally, participants may request access to the general final study findings or to published articles resulting from the study.
Supporting Information: SAP, ICF
Time Frame: Data will become available after the study results publication date and will remain accessible for up to 7 years following that date.
Access Criteria: Permission must be obtained from Universiti Teknologi Mara, the Ministry of Health Malaysia, and the Department of Orang Asli Development before access to the IPD is granted. Other researchers interested in accessing the datasets must submit a request outlining the purpose of their research. The decision to share data will be based on the reasonableness and scientific merit of the request. Access is limited strictly to anonymized IPD underlying the published study results.